CLINICAL TRIAL: NCT01664806
Title: Laparoscopic Cholecystectomy And Capacitive Coupling - Coag Versus Blend Mode and Thermal Injury to Tissue Adjacent to Port Sites
Brief Title: Laparoscopic Cholecystectomy And Capacitive Coupling - Coag Versus Blend Mode Causing Thermal Injury at Port Site Skin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 09-0049
Record Dates: First submitted 2012-08-10; First posted 2012-08-14 (Estimated); Results first posted 2013-03-01 (Estimated); Last update posted 2013-03-25 (Estimated); Status verified 2013-03

CONDITIONS: Intraoperative Complications; Thermal Injury; Electrocoagulation
Keywords: Electrosurgery; Radiofrequency energy; Monopolar instruments; Capacitive coupling; Thermal injury; Surgical complications
MeSH Terms: conditions — Intraoperative Complications; Hyperthermia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Coag mode 30 Watts Power (No Intervention): Elective laparoscopic cholecystectomy will be performed with 30 Watts power coag mode which is current standard of care.
- Covidien Triad monopolar generator (Experimental): Blend mode (triverse pencil valleylab mode) 30 Watts will be used to perform Elective laparoscopic cholecystectomy. which is the experimental arm of the study's mode.
  Interventions: Device: Covidien Triad monopolar generator

INTERVENTIONS:
Device: Covidien Triad monopolar generator — Blend mode (triverse pencil valleylab mode) 30 Watts will be used to perform a laparoscopic cholecystectomy.
  Arms: Covidien Triad monopolar generator

SUMMARY:
Monopolar radiofrequency energy is used to perform the laparoscopic cholecystectomy operation. The appearance of burns are common following laparoscopic cholecystectomy; particularly at the port site of the active electrode. Willson et al found that 9 out of 19 skin biopsies from the skin adjacent to the port site of the monopolar instrument's active electrode were found to have thermal injury by histology. [Willson et al. Surg Endosc (1997) 11:653] Authors have speculated that using different generator modes may lead to less capacitive coupling; [Wu et al Am J Surg (2000) 179: 67] although no data exists to support these speculations.

The investigators hypothesize that capacitive coupling electrosurgical injuries from monopolar instruments are occurring during laparoscopic cholecystectomy operations. The investigators hypothesize that use of blend modes will reduce the incidence of capacitive coupling thermal injuries during laparoscopic operations in comparison to coag modes.

DETAILED DESCRIPTION:
SPECIFIC AIM:

Compare incidence of skin burns caused by using coag versus blend monopolar instrument modes at the active electrode port site (epigastric port), and at the non-active electrode port sites (umbilical and right abdominal wall).

OUTCOME MEASURE:

Histologic evidence of thermal injury at the skin biopsy sites of the active electrode port, the camera port and the medial assistant port. Histology will be performed by a blinded pathologist.

POPULATION TO BE ENROLLED:

Subjects undergoing elective laparoscopic cholecystectomy will be recruited in the principle investigators pre-operative clinic. All subjects will be 18 years and older.

STUDY DESIGN AND METHODS:

Written informed consent will be obtained in all subjects prior to enrollment. Subjects will be randomized on the day of surgery to undergo the laparoscopic cholecystectomy operation with either the coag or blend modes of using standard monopolar electrosurgery instruments. The randomization process will occur by using a random number generator. A total of 40 subjects will be recruited; 20 subjects per group. Shave skin biopsies will be performed at the edge of the incisions of the active electrode port, the camera port and the medial assistant port on the right abdominal wall. The incisions and skin will be otherwise opened and closed in the routine clinical manor.

STATISTICAL ANALYSIS The incidence of skin burns created using coag or blend modes will be compared individually at all three port sites using chi-squared or Fisher's exact test where appropriate. Baseline demographic data (e.g., gender, age, body mass index, operation time, blood loss, indication for operation and histology) will be compared in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older planned to undergo elective laparoscopic cholecystectomy

Exclusion Criteria:

* Patients undergoing urgent or emergent laparoscopic cholecystectomy operations

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-11; Primary Completion 2011-08 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Robinson, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

REFERENCES:
- [Derived] Jones EL, Dunn CL, Townsend NT, Jones TS, Bruce Dunne J, Montero PN, Govekar HR, Stiegmann GV, Robinson TN. Blend mode reduces unintended thermal injury by laparoscopic monopolar instruments: a randomized controlled trial. Surg Endosc. 2013 Nov;27(11):4016-20. doi: 10.1007/s00464-013-3032-2. Epub 2013 Jun 6. PMID 23739984

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 40 patients were recruited at the University of Colorado Hospital.
Pre-assignment Details: Two screened patients were excluded because they refused entry into the trial.
Groups:
- Blend Mode (Triverse Pencil Valleylab Mode) 30 Watts: Elective laparoscopic cholecystectomy will be performed with 30 Watts power blend mode (triverse pencil valleylab mode) which is the experimental arm of the study's mode.
  Covidien Triad monopolar generator - Blend mode (triverse pencil valleylab mode) 30 Watts : Blend mode (triverse pencil valleylab mode) 30 Watts will be used to perform a laparoscopic cholecystectomy.
- Coag Mode 30 Watts Power: Elective laparoscopic cholecystectomy will be performed with 30 Watts power coag mode which is current standard of care.
  Covidien FX monopolar generator - Coag Mode 30 Watts : 30 Watts coag mode will be used to perform laparoscopic cholecystectomy
Period: Overall Study
Arm/Group | Blend Mode (Triverse Pencil Valleylab Mode) 30 Watts | Coag Mode 30 Watts Power
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Blend Mode (Triverse Pencil Valleylab Mode) 30 Watts | Coag Mode 30 Watts Power | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 19 | 37
  >=65 years | 2 | 1 | 3
Age Continuous [Mean (Standard Deviation); unit: years] | 47 (18) | 41 (12) | 44 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Histologic Thermal Injury to Epigastric Port Site Skin
Description: Shave biopsy of skin at the epigastric port site after elective laparoscopic cholecystectomy will be performed. The primary outcome is histologic evidence of burn at this port sites.
Time Frame: 1 day
Population: A sample size of convenience for feasibility.
Measure: Number; unit: participants
Arm/Group | Blend Mode (Triverse Pencil Valleylab Mode) 30 Watts | Coag Mode 30 Watts Power
Number analyzed (Participants) | 20 | 20
participants | 1 | 7

2. Secondary Outcome: Histologic Evidence of Burn at the Umbilical Port Site Skin
Description: Shave biopsy of skin at the umbilical port site after elective laparoscopic cholecystectomy will be performed. The secondary outcome is histologic evidence of burn at this port site.
Time Frame: 1 day
Population: A sample size of convenience for feasibility.
Measure: Number; unit: participants
Arm/Group | Blend Mode (Triverse Pencil Valleylab Mode) 30 Watts | Coag Mode 30 Watts Power
Number analyzed (Participants) | 20 | 20
participants | 3 | 11

ADVERSE EVENTS:
Time Frame: 1 year
Description: No adverse events were discovered.
Arm/Group | Blend Mode (Triverse Pencil Valleylab Mode) 30 Watts | Coag Mode 30 Watts Power
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
This is a pilot study with no funding so data is limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes